CLINICAL TRIAL: NCT04973709
Title: Gulhane Training and Research Hospital
Brief Title: Prevalence of Dementia and Delirium in Outpatient Clinics (DESTAN Trial)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gulhane Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Bilal Katipoglu, Principal investigator, Gulhane Training and Research Hospital
Other Study IDs: 2020-382
Record Dates: First submitted 2021-07-04; First posted 2021-07-22 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Delirium in Old Age; Delirium Superimposed on Dementia; Delirium With Dementia
Keywords: Delirium; Dementia; Mortality; Etiology; Outpatient
MeSH Terms: conditions — Delirium; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (4):
- Delirium with dementia: Delirium was detected using the short form of the Confusion Assessment Method (CAM) both at admission and daily throughout the hospital stay. Cognitive status was determined using the Mini-Mental State Exam, Clinical Dementia Rating (CDR). Dementia was defined by a CDR score of 1. The primary independent variable was a composite of delirium and dementia diagnosis, and we examined the overlap by categorizing the cases into four groups: no delirium or dementia, dementia alone, delirium alone, and DSD.
  Interventions: Diagnostic Test: Confussion assessment method (CAM); Diagnostic Test: Dementia diagnosis
- Dementia without Delirium: Delirium was detected using the short form of the Confusion Assessment Method (CAM) both at admission and daily throughout the hospital stay. Cognitive status was determined using the Mini-Mental State Exam, Clinical Dementia Rating (CDR). Dementia was defined by a CDR score of 1. The primary independent variable was a composite of delirium and dementia diagnosis, and we examined the overlap by categorizing the cases into four groups: no delirium or dementia, dementia alone, delirium alone, and DSD.
  Interventions: Diagnostic Test: Dementia diagnosis
- Delirium without Dementia: Delirium was detected using the short form of the Confusion Assessment Method (CAM) both at admission and daily throughout the hospital stay. Cognitive status was determined using the Mini-Mental State Exam, Clinical Dementia Rating (CDR). Dementia was defined by a CDR score of 1. The primary independent variable was a composite of delirium and dementia diagnosis, and we examined the overlap by categorizing the cases into four groups: no delirium or dementia, dementia alone, delirium alone, and DSD.
  Interventions: Diagnostic Test: Confussion assessment method (CAM)
- No dementia, No delirium: Delirium was detected using the short form of the Confusion Assessment Method (CAM) both at admission and daily throughout the hospital stay. Cognitive status was determined using the Mini-Mental State Exam, Clinical Dementia Rating (CDR). Dementia was defined by a CDR score of 1. The primary independent variable was a composite of delirium and dementia diagnosis, and we examined the overlap by categorizing the cases into four groups: no delirium or dementia, dementia alone, delirium alone, and DSD.

INTERVENTIONS:
Diagnostic Test: Confussion assessment method (CAM) — Participants enrolled in the Delirium group according to the CAM.
  Groups: Delirium with dementia; Delirium without Dementia
Diagnostic Test: Dementia diagnosis — Participants enrolled in the Dementia group according to the CDR scores and MMSE scores and DSM4/5 criteria
  Groups: Delirium with dementia; Dementia without Delirium

SUMMARY:
The aim of this study is to assess the prevalence and etiologic risk factors of delirium in outpatient geriatric patients and also hospitalized patients.

DETAILED DESCRIPTION:
This study aimed to investigate the frequency of delirium and examines the association between delirium and other possible risk factors and prognostic factors (dementia etc.)

ELIGIBILITY:
Inclusion Criteria:

* We included all 65 years older patients who evaluated according to a comprehensive geriatric assessment that is consistently performed during admission to the outpatients' clinic of the hospital.

Exclusion Criteria:

* Exclusion criteria were serious psychiatric disorders such as schizophrenia or major depression.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Community-dwelling older adults (65 years and older)
Sampling Method: Non-Probability Sample
Enrollment: 714 (Estimated)
Dates: Start 2021-08-05 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2025-11-11 (Estimated)

PRIMARY OUTCOMES:
frequency of Mortality | 1 year fellow-up
  1st year mortality according to the electronic national data base

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Naharcı, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Gulhane training and research hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Katipoglu B, Demircan SK, Naharci MI. Association of drug burden index with delirium in community-dwelling older adults with dementia: a longitudinal observational study. Int J Clin Pharm. 2023 Oct;45(5):1267-1276. doi: 10.1007/s11096-023-01551-7. Epub 2023 Mar 18. PMID 36933080